| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

# **Revision History**

| Revision | Revision Date | Reason for Revision/Change Request | Revised By |
|---|---|---|---|
| 1.0 | 14-March-2018 | Original Release | Daniel Manas, DMS |
| 2.0 | 14-Nov-2018 | Updated version | Daniel Manas, DMS |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

# Final Statistical Analysis Plan

A Double Blind, Randomized, Placebo Controlled, Dose Escalation Phase 2a Clinical Trial for the Evaluation of Safety and Thermogenesis-induction of RZL-012 in Overweight and Obese Volunteers





# TABLE OF CONTENTS

| l. | DEFINITIONS AND/OR ABBREVIATIONS | 4 |
|----|----------------------------------|----|
| 2. | PURPOSE | 10 |
| 3. | SCOPE | 10 |
| 4. | RESPONSIBILITIES | 11 |
| 5. | PROCEDURE | 12 |
| 6. | RELATED DOCUMENTS (optional) | 27 |
| 7. | RELATED FORMS (optional) | 27 |
| 8. | REFERENCES | 28 |
| 9. | Appendices (optional) | 28 |
| | 9.1 APPENDIX I: TABLE SHELLS | 28 |
| | 9.2 APPENDIX II: LISTINGS SHELLS | 30 |



# SIGNATURES PAGE

| Daniel Manas, author | |
|-----------------------------------------|-------|
| Senior Biostatistician & SAS programmer | |
| MediStat Ltd. | Date: |
| Daphna Goffer, reviewer | |
| Senior Biostatistician & SAS programmer | |
| MediStat Ltd. | Date: |
| Rachel Gueta | |
| Raziel Therapy Ltd. | Date: |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

# 1. DEFINITIONS AND/OR ABBREVIATIONS

| ADR | Adverse drug reaction |
|------------------|-----------------------------------------|
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| ATP | Adenosine triphosphate |
| AUC | Area under the concentration-time curve |
| BAT | Brown-like adipose tissue |
| BMI | Body Mass Index |
| BUN | Blood urea nitrogen |
| °C | Degrees Celsius |
| CBC | Complete blood count |
| CDC | Center for Disease Control |
| cGMP | Current Good Manufacturing Practices |
| CI | Confidence Interval |
| CK-MM | Creatine Kinase - Muscle |
| C <sub>max</sub> | Maximum observed concentration |
| CNS | Clinically not significant |
| CRF | Case Report Form |
| CPK | Creatine phosphokinase |
| CRP | C-reactive protein |

| Medi-Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

| CS | Clinically significant |
|------------------|------------------------------------------------|
| СТС | Common terminology criteria |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DICOM | Digital Imaging and Communications in Medicine |
| DSMB | Data and Safety Monitoring Board |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| EF | Efficacy analysis set |
| ER | Emergency room |
| FDA | Food and Drug Administration |
| FFA | Free fatty acids |
| FIFO | First In First Out |
| FLASH | Fast-low-angle shot |
| FOB | Functional Observational Battery |
| GLP | Good Laboratory Practice |
| GTTP | Gamma-glutamyltransferase |
| HBV | Hepatitis B virus |
| HCRC | Hadassah Clinical Research Center |
| HCV | Hepatitis C virus |
| H&E | Hematoxylin and eosin stain |
| HDL | High-density lipoprotein |
| HED | Human equivalent dose |
| HIV | Human immunodeficiency virus |
| IC <sub>50</sub> | Half maximal inhibitory concentration |



| ICF | Informed Consent Form |
|---|---|
| ICH-GCP | International Conference on Harmonization Good Clinical Practice |
| IFN | Interferon |
| IL | Interleukin |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| LDL | Low-density lipoprotein |
| LDH | Lactate dehydrogenase |
| LPL | Lipoprotein lipase |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCP | Monocyte chemoattractant protein |
| MCV | Mean corpuscular volume |
| MD | Medical Doctor |
| MEDDRA | Medical Dictionary for Regulatory Activities |
| | , , , |
| NOAEL | No observed adverse effect level |
| NSAIDs | Non Steroid Anti-Inflammatory Drugs |
| Pl | Principal Investigator |
| PK | Pharmacokinetics |
| PKA | PK Analysis set |
| PT | Prothrombin time |
| MEDDRA MPV MRI NHANES NOAEL NSAIDs PI PK PKA | Medical Dictionary for Regulatory Activities Mean platelet volume Magnetic Resonance Imaging National Health and Nutrition Examination Survey No observed adverse effect level Non Steroid Anti-Inflammatory Drugs Principal Investigator Pharmacokinetics PK Analysis set |

| Medi-Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

| PTT | Partial thromboplastin time |
|------------------|-----------------------------------------------|
| QA | Quality Assurance |
| RBC | Red blood cells |
| RDW | Red cell distribution width |
| SA | Safety analysis set |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SAT | Subcutaneous adipose tissue |
| SC | Subcutaneous |
| SFM | Subcutaneous fat mass |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| T <sub>1/2</sub> | Terminal half-life |
| TAG | Triacylglycerols |
| TBD | To be determined |
| TC | Total Cholesterol |
| TG | Triglycerides |
| TGF | Transforming growth factor |
| T <sub>max</sub> | Time of maximum observed sample concentration |
| TNF | Tumor necrosis factor |
| UCP1 | Uncoupling protein 1 |
| ULN | Upper limit of normal |
| US/USA | United States/United States of America |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

| WAT | White adipose tissue |
|-----|---------------------------|
| WBC | White blood cells |
| WHO | World health organization |
| WHR | Waist to hip ratio |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

## 2. PURPOSE

- 2.1 The purpose of this document is to describe in detail the Statistical Analysis Plan of clinical study procedures carried out by Medistat Ltd.
- 2.2 This document serves Medistat Ltd. as a guiding document for all statistical analyses performed at the end of each clinical study.
- 2.3 This SAP is specific to Raziel Therapeutics LTD, study RZL-012-P2aUS-001.4
- 2.4 This SAP aims to provide details on: sample size calculation, efficacy analyses and safety analyses.

## 3. SCOPE

- 3.1 This document applies to all members of the statistical & data management units in Medistat Ltd.
- 3.2 This document includes the main and interim study trial analysis.

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

## 4. RESPONSIBILITIES

# 4.1 Medistat Ltd. Responsibilities

The following personnel are responsible for these activities:

| Activities | Responsible and | Title |
|---|---|---|
| | accountable | |
| Statistical Analysis Plan | Daniel Manas | Senior Biostatistician |
| (SAP) | | & SAS Programmer |
| Statistical Report and listing | Daniel Manas | Senior Biostatistician |
| appendix | | & SAS Programmer |
| Quality Assurance (QA) of | David Israel | Senior Biostatistician |
| SAP and programs | | & SAS Programmer |
| Quality Assurance (QA) of | Shimrit Herbst | Quality & Data |
| final report | | Assurance Manager |

# 4.2 Raziel's Responsibilities

- 4.2.1 To review and approve the SAP and related documents prior to database lock.
- 4.2.2 To review and approve the draft and final statistical report and listing appendix.

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

#### 5. PROCEDURE

#### 5.1 Introduction

- 5.1.1 This Statistical Analysis Plan (SAP) is based on the study protocol final version V1.4, dated 4 March, 2018.
- 5.1.2 This Statistical Analysis Plan (SAP) contains details of the statistical analyses that will be performed, providing a more detailed description of the approach defined in the study protocol. Definitions of variables and populations used for the analyses are also included. The SAP will be finalized and signed prior to hard lock of the database.
- 5.1.3 General output specifications are provided; examples are given of calculations of derived variables.

#### 5.2 Rationale

- 5.2.1 The purpose of this study is to test safety and efficacy of a new chemical entity, RZL-012, in converting WAT into a thermogenic tissue and reducing fat-mass in overweight and obese males
- 5.2.2 RZL-012 investigational drug is intended for a single dose in multiple injections into the subcutaneous fat. The injection dosing regimen and technique is crucial for the therapy safety and efficacy. The RZL-012 drug is a ready to use liquid to be injected to the subcutaneous fat, supplied in a 1 vial kit. 1 vial contains 250 mg/4.8 mL RZL-012 in formulation F12. The vehicle is a ready to use liquid to be injected to the subcutaneous fat, supplied in a 1 vial kit. 1 vial contains 4.8 mL of formulation F12.

## 5.3 Study Objectives and Endpoints

- 5.3.1 Primary Objectives:
- 5.3.2 Evaluation of the overall safety and preliminary efficacy of RZL-012 after injection into the subcutaneous fat.
- 5.3.3 Primary Endpoints



- 5.3.4 Safety: The main objective is the evaluation of the overall safety of RZL-012 injection into the subcutaneous fat. Therefore, the primary endpoint will be the incidence of intolerable side effects and all adverse events of RZL-012 injection into the subcutaneous fat. The dose escalation scheme will be stopped if at any dose cohort, 2 patients will experience intolerable side effects.
- 5.3.5 Efficacy: The primary endpoint for efficacy is a significant thermogenesis at the injected site compared with the contra-lateral, non-injected site. This was monitored by sensitive (± 0.1 °C) Infra-Red thermal camera. A thermogenic effect is defined by an increase of 1 °C in the injected site when compared to the surroundings and/or the non-injected site, apparent at least 28 days after injection and non-related to inflammatory response as determined by inflammatory cytokines. The primary efficacy evaluation will be supported by results from secondary endpoints, including MRI, biopsy and biomarkers
- 5.3.6 Secondary Objectives:
- 5.3.7 Determination of RZL-012 pharmacodynamics and pharmacokinetics. Evaluation of the existence of a thermogenic effect and the extent, duration and tissue associated changes of the thermogenic response to RZL-012, via minimal invasive means (injected-site thermogenesis imaging, Magnetic Resonance Imaging (MRI) and biopsy) after subcutaneous injection into fatty tissue below the skin.
- 5.3.8 Secondary Endpoints
- 5.3.9 Duration of the thermogenic effect, defined as a net-delta  $\geq 1$
- 5.3.10 Local reduction in fat mass as determined by MRI.
- 5.3.11 Clinical laboratory changes from baseline including improvement in fasting blood glucose and lipid profile.
- 5.3.12 Establishing pharmacokinetic profile for RZL-012.
- 5.3.13 Anthropometric changes from baseline, including body weight change.
- 5.3.14 Elucidation of the histological changes account for the thermogenic effect by biopsy of the injection site.
- 5.3.15 Change from baseline in inflammatory markers and cytokines.
- 5.4 Overall study design and plan

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

- 5.4.1 Study Design
- 5.4.2 This is a consecutive 4 cohort, dose escalation placebo-controlled clinical trial in overweight and obese subjects. All cohorts will be comprised of 6 active (RZL-012) and 2 placebo subjects.
- 5.4.3 Within each cohort, dosing of the first 3 subjects will progress consecutively from one individual to the other at 7-day intervals. For additional precaution, the first 3 subjects will be forced randomized into 2 active and 1 control. This study design will allow the physicians to monitor safety in a two subjects at each dose, nevertheless the blindness will remain intact. The remaining subjects in a cohort will be randomized to either active treatment or placebo in a ratio determined by the number of subjects targeted for each cohort. Dosing of the next subjects will be in couples and the last subjects will be in a triplet.

## 5.4.4 Schedule of Assessments

| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Visit Schedule (Days 1 to 28) | | | | | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>(Days<br>29 -<br>168) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| Signed informed consent | X | | | | | | | | | | |
| Medical<br>history | X | | X | | | | | | | | |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018 REVISION NUMBER: 2.0 |

| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Vi | Visit Schedule (Days 1 to 28) | | | | | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>1 (Days<br>29 -<br>168) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| Complete physical exam | X | | | | | | | | | X | |
| Serology<br>assays (HBV,<br>HCV, HIV) | X | | | | | | | | | | |
| Fasting glucose | X | | X | | | | | | | | |
| Fasting glucose, insulin, leptin and lipid profile (including FFA) | | | X | | | | | | | X | Every<br>28 days |
| Inflammatory markers and Cytokines - In subject of the 2 <sup>nd</sup> , 3 <sup>rd</sup> and 4 <sup>th</sup> cohorts <sup>b</sup> | | | X | | | | X | X | X | X | |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Visit Schedule (Days 1 to 28) | | | | | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>(Days<br>29 -<br>168) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| Photography<br>of site of<br>injection and<br>contralateral | X | | | | X | | X | X | X | X | Every<br>28 days |
| MRI section around the umbilicus | | X | | | | | | | | X | |
| MRI section<br>around the<br>umbilicus – for<br>cohort 2 | | | | | | | | | | | On Day |



| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Vi | isit Scl | nedule | (Days | s 1 to 2 | :8) | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>1 (Days<br>29 -<br>168) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| MRI section around the umbilicus – for 3 <sup>rd</sup> and 4 <sup>th</sup> cohort or in cohort 2 if 2 subject experience intolerable side effects in cohort 3) | | | | | | | | | | | Every<br>28 days |
| Anthropometri c measurements: (weight, height) BMI, (waist & hip circumference) WHR | X | X | X | | | | | | | X | Every<br>28 days |
| Weight – by<br>the subjects at<br>home – | | | | | | | X | X | X | | On<br>weeks<br>when |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018 REVISION NUMBER: 2.0 |

| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Visit Schedule (Days 1 to 28) | | | 8) | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>(Days<br>29 -<br>168) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| morning(8-<br>12hr overnight<br>fast) and<br>evening | | | | | | | | | | | not<br>visiting<br>the site |
| Urine Drug<br>Screen | X | | X | | | | | | | | |
| Infra-Red<br>thermal<br>imaging of the<br>injected site | X | | X | | X | | X | X | X | X | On Day |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018 REVISION NUMBER: 2.0 |

| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Vi | isit Scl | nedule | (Days | s 1 to 2 | 8) | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>1 (Days<br>29 -<br>168) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| Infra-Red thermal imaging of the injected site - for 3 <sup>rd</sup> and 4 <sup>th</sup> cohort or in cohort 2 if 2 subjects experience intolerable side effects will in cohort 3) <sup>k</sup> | | | | | | | | | | | Every<br>28 days |
| Serum<br>Chemistry,<br>Hematology <sup>c</sup> | X | | X | | X | X | X | X | | X | |
| Histamine levels <sup>d</sup> | | | X | | X | X | | X | | | |
| Urinalysis Pharmacokinet ics f | X | | | Pre <sup>e</sup> X post <sup>e</sup> | X | | | X | | X | |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Visit Schedule (Days 1 to 28) | | | (8) | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts 1 (Days<br>29 -<br>168) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| Draize score at the injected site <sup>g</sup> | X | | | Pre <sup>e</sup> X<br>post <sup>e</sup> | X | | X | X | X | X | Every<br>28 days |
| Vital signs h | X | | | Pre <sup>e</sup> X post <sup>e</sup> | X | | X | X | X | X | |
| Injection of RZL-012 | | | | X | | | | | | | |
| ECG i | X | | | X post e | X | | | X | | X | |
| Pulse rate <sup>j</sup> | | | | Pre <sup>e</sup> X post <sup>e</sup> | X | | | | | | |
| Adverse event assessment | | | | | X | | | | <b>→</b> | | Every<br>28 days |
| Adverse event assessment by phone for cohorts 1 and 2 | | | | | | | | | | | On Day<br>84 and<br>112 |



| Study<br>Procedure | Screening<br>Day 1 | Screeni<br>ng Day<br>2 | Clinic<br>Admissi<br>on | Baseline<br>(Treatme<br>nt) | Visit Schedule (Days 1 to 28) | | | 28) | Follow-<br>up<br>Schedu<br>le for<br>the<br>highest<br>dose<br>cohorts<br>(Days<br>29 -<br>168) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-<br>28)<br>throug<br>h Day<br>(-7) | Day <sup>a</sup> -(-<br>14)<br>through<br>Day (-2) | Day (-1) | Day <sup>a</sup> 0 | Da<br>y 1 | Da<br>y 3 | Da<br>y 7 | Day<br>14 | Da<br>y<br>21 | Da<br>y<br>28 | Day 56,<br>84, 112,<br>140,<br>168 |
| Subjects diary recording weight | | | | | | | X | X | X | | On weeks when not visiting the site |
| Biopsy – In subject of cohort 3 (or in cohort 2 if 2 subjects experience intolerable side effects in cohort 3) <sup>k,l</sup> | | | | | | | | | | | On Day<br>56 |

- a. Study day is based on Day 0 defined as the day of RZL-012 injection.
- b. Inflammatory markers and cytokines from the 2<sup>nd</sup>, 3<sup>rd</sup> and 4<sup>th</sup> cohorts (on 6 RZL-012 treated and 2 placebo treated subjects in each cohort): CRP, Adiponectin, CD-163, Interleukin [IL]-1β, IL-4, IL-6, IL-10, IL12p70, IL-13, IL-23, Tumor necrosis factor [TNF] α and TGFβ1.
- CBC, coagulation, serum chemistry analysis, renal and liver function, urinalysis, CPK, amylase measurement: before injection, 14d and 28d following injection
- d. Histamine blood level measurement: clinical admission, following drug injection (24h ± 2h), 3d and 14d following injection
- e. Pre/post refers to before/after injection respectively
- f. Pharmacokinetics at the given time points: 0, 30, 60 min, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 30h in subjects from the 1<sup>st</sup>, 2<sup>nd</sup> and 3<sup>rd</sup> cohorts. Pharmacokinetics will not be conducted in the fourth cohort as the injected dose is divided in 2 clusters 2 weeks apart.

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

- g. Draize score evaluation: before injection, 2h, 24h and 7d,14d,21d and 28d following injection
- h. Vital signs measurement: before injection, 2h, 24h and 7d,14d,21d and 28d following injection
- i. ECG is to be performed in triplicate for all measurements in given time point: 4h, 12h, 24h, Day 14 and 28 following injection
- j. Pulse rate measurements at given time points: 1h, 2h, 4h, 8h, 12h, 24h following injection in the opposite hand of blood sampling
- k. For 3 subjects of cohort 3 (in cohort 2 if 2 subjects experience intolerable side effects in cohort 3) if thermogenesis is evident by thermal camera by Day 56, biopsy from the injected for histology and BAT characterization.
- 1. For subjects from the 3rd (or in cohort 2 if 2 subjects will experience intolerable side effects within the 3rd cohort) and 4th cohort

| Medi-Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

- 5.4.5 Randomization, Blinding and Un-blinding
- 5.4.6 Subjects will be randomized to each study group, i.e., investigational therapy or control, left side injection or right side injection according to a predefined randomization scheme. The investigational therapy group will be treated with RZL-012 and the control group will be treated with the same formulation (vehicle) as with RZL-012, absent active medication
- 5.4.7 Masking will be used to blind the Investigator regarding randomization, i.e., assignment to study group will be disclosed only after subject eligibility is confirmed and immediately before treatment initiation. The pharmacist will be unmasked and will be responsible to fill the syringes for injection.
- 5.5 Selection of study population
  - 5.5.1 Study Population
  - 5.5.2 Male subjects
  - 5.5.3 Age 20 60 years old
  - 5.5.4 The study population include subjects who are obese by Body Mass Index (BMI) definition (27.5 < BMI ≤ 34.9)
  - 5.5.5 Rationale Sample Size Calculation
  - 5.5.6 The planned sample size is 32 subjects (8 in each cohort). 6 subjects per dose group paradigm with the addition of a 2 subjects per control group for all doses. A maximum of 32 evaluable subjects will be included in the study (24 in the RZL-012 treatment arm and 8 in the placebo arm) and followed for as long as 3 months in the 2 lowest dose cohorts, and in the 2 highest dose cohorts for up to 5 months.
- 5.6 Statistical Analysis Software and Data Management
  - 5.6.1 Data manipulation, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed using SAS® version 9.3 or higher for Windows. If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.
  - 5.6.2 Data Management
  - 5.6.3 Data management for the study is performed by Spaulding Clinical.
  - 5.6.4 Medical Coding



- 5.6.5 Concomitant medications entered into the database are coded using the WHO (World Health Organization) Drug Public Website Dictionary named WHOCC-ATC/DDD index, which employs the Anatomical Therapeutic Chemical classification system.
- 5.6.6 Adverse events are coded using the most updated version of Medical Dictionary for Regulatory Activities (MedDRA) terminology.
- 5.6.7 Medical history events are coded using the most updated version of Medical Dictionary for Regulatory Activities (MedDRA) terminology
- 5.6.8 Handling of Missing data
- 5.6.9 No imputation of missing data will be performed
- 5.6.10 Protocol Violations and Deviations
- 5.6.11 Departures from the protocol should be avoided unless required for the safety of the subject. Protocol deviations and, if possible, the reason for occurrence will be documented by the study monitor and included in the final clinical study report.
- 5.6.12 The Investigator must report any protocol deviation to the Sponsor and, if required, to the IRB/IEC in accordance with local regulations, within reasonable time. All violations and deviations must be recorded in the study site's electronic system and signed by the Investigator (or designee).

#### 5.7 Subject Population for analyses

- 5.7.1 The safety analysis set (SA) will consist of all enrolled subjects who received the study treatment, either RZL-012 or placebo (exposed population), including subjects prematurely withdrawn. All enrolled subjects receiving at least one study drug injection are considered evaluable for the SA set.
- 5.7.2 The SA analysis set will serve as the principal data analysis set for the analyses of the safety endpoints.
- 5.7.3 The efficacy analysis set (EF) will consist of all subjects from the SA analysis set without any major protocol violations measured at baseline
- 5.7.4 The EF analysis set will serve as the principal data analysis set for the analyses of the efficacy endpoints.

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

- 5.7.5 The PK analysis set will consist of all subjects with no major deviations related to study drug administration (e.g., incomplete injection of study drug).
- 5.7.6 The PK analysis set will serve as the principal data analysis set for the PK analysis

## 5.8 Statistical Analysis

- 5.8.1 General
- 5.8.2 All measured variables and derived parameters will be listed individually and, if appropriate, tabulated by descriptive statistics. For categorical variables summary tables will be provided giving sample size, absolute and relative frequency. For continuous variables summary tables will be provided giving sample size, arithmetic mean, standard deviation, standard error, coefficient of variation (CV%), median, minimum and maximum of variables, and 95% confidence intervals of means.
- 5.8.3 The data is analyzed using the SAS ® version 9.3 or higher (SAS Institute, Cary North Carolina). Analyses presented in the clinical report but not mentioned in the SAP are unplanned or ad-hoc analyses.
- 5.8.4 Statistical methods presented in the SAP may be slightly different from those that are presented in the protocol. Differences are clearly stated and the SAP supersedes the protocol only with regard to the way data will be handled and analysed.
- 5.8.5 Derived Data
- 5.8.6 Definition of baseline
- 5.8.7 Baseline is defined as the last non-missing value prior to the patient start of treatment (screening or baseline visit).
- 5.8.8 End of Study
- 5.8.9 The end-of-study visit is defined as Day 168.
- 5.8.10 Disposition of subjects (Table 14.1-1 14.1.2)
- 5.8.11 The number of subjects that are randomized into the study, the number of subjects in the Safety, efficacy analysis set, and PK populations, and the number of study completers will be presented.
- 5.8.12 The reasons for early termination/ withdrawal will be summarized.



- 5.8.13 Demographic and Baseline data (Tables 14.1-3-14.1-4)
- 5.8.14 Baseline and demographic data will be summarized in appropriate tables using the Safety population. The data includes demographic characteristics (age and gender) and medical history.
- 5.8.15 Efficacy Analysis
- 5.8.1 The primary endpoint for efficacy is a significant thermogenesis at the injected site compared with the contra-lateral, non-injected site.
- 5.8.2 The average temperature will be presented in a tabular form by visit, side (treated / not treated) and treatment received (RZL-012 / placebo) by cohort and overall. Difference between the sides (treated not treated) will be presented in a tabular form by visit treatment along with the change from baseline (net-delta) in these differences by cohort and overall.
- 5.8.3 Kruskal-Wallis will be used to compare the net-delta between the study arms for the relevant cohorts and visits.
- 5.8.4 The number and percent of subjects with a thermogenic effect, defined as a net-delta ≥ 1, will be presented by cohort and visit for the subjects in the active arm. The duration of the thermogenic effect after the Day 28 visit, for subjects in the active arm with thermogenic effect at the Day 28 visit will be presented.
- 5.8.5 Subcutaneous Fat Mass (SFM) ratio (treated sites / control sites) averaged over the MRI slices will be presented in tabular form by visit, treatment and cohort. The change from baseline in this ratio (in % from the ratio at baseline) will be presented in the same manner, and compared between the treatment arms with Kruskal-Wallis test.
- 5.8.6 Changes from baseline in fasting blood glucose, lipid profile, anthropometric changes, inflammatory markers and cytokines will be presented by visit, treatment, and cohort.
- 5.8.7 Histology results will be presented in tabular form by treatment for relevant subjects.
- 5.8.8 Safety analysis
- 5.8.9 Safety data will be summarized for the Safety population.
- 5.8.10 Adverse events will be coded according to coding dictionaries (the most updated version of MedDRA) and presented in tables by System Organ Class (SOC) and Preferred Term (PT) and by treatment group.



- 5.8.11 The incidence of AEs, as well as the intensity and relationship to study drug will be summarized by treatment group.
- 5.8.12 The incidence of all adverse events will be presented by treatment overall and by cohort along with two sided 95% exact binomial Confidence Interval (CI).
- 5.8.13 The incidence of intolerable side effects will be presented by treatment overall and by cohort along with two sided 95% exact binomial Confidence Interval (CI).
- 5.8.14 Concomitant medication verbatim terms (as recorded on the CRFs) will be coded to Anatomical Therapeutic Chemical (ATC) Level 2 and 4 using the World Health Organization (WHO) dictionary.
- 5.8.15 Interim Analysis
- 5.8.16 An interim analysis is planned at the end of each cohort for evaluation of efficacy. For this purpose, a data lock (except for externally collected data such as PK) will be implemented after each cohort is completed. Upon lack of trends in efficacy due to effect size, the Sponsor will consider study termination

# 6. RELATED DOCUMENTS (OPTIONAL)

- 6.1 Study Protocol: RZL-012-P2aUS-001.4\_track changes 04 Mrch 2018
- 6.2 Randomization plan: RZL-012-P2aUS random plan final version 1.0 01-08-2017.pdf

## 7. RELATED FORMS (OPTIONAL)

Not Applicable

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

#### 8. REFERENCES

Not Applicable

## 9. APPENDICES (OPTIONAL)

9.1 APPENDIX I: TABLE SHELLS

14.1 Demographic Data

Table 14.1-1: Disposition of Subjects

Table 14.1-2: Analysis populations

Table 14.1-3: Demographic Data

Table 14.1-4: Medical History

14.2 Efficacy Assessment

14.2.1 Primary Safety Endpoint

Table 14.2.1-1: Summary of Thermal Imaging per visit

Table 14.2.1-2: Summary of Thermal Imaging Changes per visit

P-value for difference between groups

Table 14.2.1-3: Frequency of Thermogenic Effect

Table 14.2.1-4: Duration of Thermogenic Effect

Table 14.2.1-5: Summary of MRI Results

14.2.2 PK Assessments

Table 14.2.2-1: Summary Statistics of RZL-012 Concentrations (ng/mL) by Treatment and time (hours)

Table 14.2.2-2: Summary of RZL-012 PK Parameters by Treatment

14.3 Safety Data

14.3.1 Adverse Events

Table 14.3.1-1: Frequency of Any Adverse Events

Table 14.3.1-2: Frequency of any intolerable side effects

Table 14.3.1-3: Summary of Adverse Events by SOC and PT by treatment

Table 14.3.1-4: Summary of Adverse Events by SOC, PT, severity, and by treatment

14.3.2 Other safety Assessments

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

Table 14.3.2-1: Summary of Vital signs

Table 14.3.2-2: Changes from baseline - Vital signs

Table 14.3.2-3: Summary of Chemistry

Table 14.3.2-4: Changes from baseline – Chemistry

Table 14.3.2-5: Summary of Hematology

Table 14.3.2-6: Changes from baseline – Hematology

Table 14.3.2-7: Summary of Coagulation

Table 14.3.2-8: Changes from baseline – Coagulation

Table 14.3.2-9: Summary of Glucose

Table 14.3.2-10: Changes from baseline - Glucose

Table 14.3.2-11: Summary of Lipids

Table 14.3.2-12: Changes from baseline - Lipids

Table 14.3.2-13: Summary of Plasma

Table 14.3.2-14: Changes from baseline - Plasma

Table 14.3.2-15: Summary of Serum

Table 14.3.2-16: Changes from baseline – Serum

Table 14.3.2-17: Summary of Urinalysis

Table 14.3.2-18: Changes from baseline - Urinalysis

Table 14.3.2-19: Summary of Urinalysis - Categorical results

Table 14.3.2-20: Summary of Serology at Screening

Table 14.3.2-21: Summary of Drug Screening

Table 14.3.2-22: Summary of ECG Results

Table 14.3.2-23: Changes from baseline - Urinalysis

Table 14.3.2-24: Summary of Draize Score

Table 14.3.2-25: Summary of Physical Examination

Table 14.3.2-26: Any concomitant medications

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

9.2 APPENDIX II: LISTINGS SHELLS

16.2.1 Subject Disposition

Listing 16.2.1-1: Subject Disposition

Listing 16.2.1-2: Visit dates per subject

16.2.2 Protocol Deviations

Listing 16.2.2-1: Inclusion/Exclusion Criteria

16.2.3 Subjects Excluded from the Efficacy Analysis

Listing 16.2.3-1: Subjects Excluded from the Efficacy and PK Analysis

16.2.4 Demographic Data and Baseline Assessments

Listing 16.2.4-1: Demographic Data

Listing 16.2.4-2: Medical History

16.2.5 Compliance/Exposure/Drug Concentration Data

Listing 16.2.5-1: Index Procedure

16.2.6 Individual Efficacy/PK/PD Response Data

Listing 16.2.6-1: PK Collection

Listing 16.2.6-2: Thermogenesis results

Listing 16.2.6-2: RZL-012 Concentration (ng/mL) by Subject, Treatment and Time

Listing 16.2.6-3: RZL-012 PK Parameters by subject and Treatment

Listing 16.2.6-5: MRI results

16.2.7 Adverse Events

Listing 16.2.7-1: Adverse Events

16.2.8 Laboratory and other safety parameters

Listing 16.2.8-1: Chemistry

Listing 16.2.8-2: Hematology

Listing 16.2.8-3: Coagulation

Listing 16.2.8-4: Urinalysis

Listing 16.2.8-5: CK, Total+Isoenzymes, and Serum

Listing 16.2.8-6: Plasma

Listing 16.2.8-7: Glucose

Listing 16.2.8-8: Lipids

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | | EFFECTIVE DATE: 14/Nov/2018<br>REVISION NUMBER: 2.0 |

Listing 16.2.8-9: Drugs of Abuse

Listing 16.2.8-10: Serology

Listing 16.2.8-11: Vital Signs

Listing 16.2.8-12: ECG Findings

Listing 16.2.8-13: ECG Quantitative Results

Listing 16.2.8-14: Abnormal Physical Examination

Listing 16.2.8-15: Draize Assessment

Listing 16.2.8-16: Concomitant Medications